CLINICAL TRIAL: NCT04171011
Title: Feasibility of Splenic Nerve Stimulation During Esophagectomy
Brief Title: Nerve Stimulation During Esophagectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galvani Bioelectronics (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: GAL1018
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Inflammatory Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nerve Stimulation (Experimental): Participants will undergo brief NVB stimulation during the esophagectomy procedure.
  Interventions: Device: Stimulator device

INTERVENTIONS:
Device: Stimulator device — The stimulator device will be used to electrically stimulate the NVB

SUMMARY:
Esophagectomy is the cornerstone for treatment of esophageal cancer. However, it is associated with substantial morbidity and mortality. Studies suggest that systemic inflammation after surgery has a negative impact on surgical outcomes. Attenuation of an excessive inflammatory response within the perioperative period for high-risk surgical procedures may reduce morbidity and mortality. The inflammatory response may be important in the development of these complications and reduction of inflammatory cytokine may be associated with an improved outcome.

The current study will evaluate the feasibility and safety of neuromodulation during minimally invasive surgery for esophageal cancer (esophagectomy) to assess impact on the inflammatory response. During the esophagectomy, a stimulation lead will be placed on the exposed nerves, and energy applied to the lead to test whether the nerves can be activated. The study will also measure potential physiological responses to nerve activation.

DETAILED DESCRIPTION:
Active dampening of the inflammatory response may be an important therapeutic target to decrease complications and improve recovery following esophagectomy. The current study is intended to evaluate the feasibility and safety of stimulating the exposed nerves in esophagectomy patients.

During minimally invasive esophagectomy, a neurovascular bundle (NVB) is exposed or partially exposed as part of the obligatory lymph node dissection. At the point in the esophagectomy when the NVB is being isolated, a lead will be applied laparoscopically to the NVB and connected to an external pulse generator. An ultrasound transducer will be introduced to the abdomen and placed on the NVB to visualize splenic arterial blood flow. The NVB will be stimulated while physiologic responses are observed. Blood samples will be taken before, and at certain pre-defined time points after, stimulation and recovery. The lead and ultrasound transducer will be removed after completion of stimulation, and the esophagectomy surgery will continue. Surgeon experience applying and removing the cuff electrode will be documented, in addition to the responses to NVB stimulation. Post-operative safety will be followed through 7-days (or day of discharge if earlier).

ELIGIBILITY:
Inclusion Criteria:

* Female of non-reproductive potential or male
* Undergoing minimally invasive esophagectomy
* Confirmed presence of splenic NVB loop via imaging prior to surgery
* Age equal or above 21 years at the screening visit
* Capable of giving signed informed consent (IC)
* Normal blood pressure, or hypertensive managed with medication such that they are deemed fit for surgery

Exclusion Criteria:

* Previous splenectomy
* Existing implantable device
* Active pancreatitis or history of severe pancreatitis with complications, hepatic or splenic disease
* Use of oral steroids 4 weeks prior to inclusion
* Current use immunosuppressive agents or biologicals. Previous use of biologicals is allowed, if a washout period of 2 months is applied
* Use of anticoagulants within 1 week of surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Feasibility applying and removing the stimulation lead: Proportion of participants in whom the lead was successfully applied and removed | 1 day
  Proportion of participants in whom the lead was successfully applied and removed
Safety of placement, stimulation and removal of the lead: Incidence of adverse events | 7 days
  Incidence of adverse events

SECONDARY OUTCOMES:
Peak Systolic Velocity (PSV) blood flow change measured by doppler ultrasound | Before stimulation and during stimulation
End Diastolic Velocity (EDV) blood flow change measured by doppler ultrasound | Before stimulation and during stimulation
Velocity Time Integral (VTI) blood flow change measured by doppler ultrasound | Before stimulation and during stimulation

OTHER OUTCOMES:
Heart Rate (HR) change | Before stimulation and during stimulation
Systolic Blood Pressure (SBP) change | Before stimulation and during stimulation
Diastolic Blood Pressure (DBP) change | Before stimulation and during stimulation
Mean Arterial Blood Pressure (MAP) change | Before stimulation and during stimulation
Hematology (white blood cell (WBC) counts) | Before stimulation to Day 1 post stimulation
Cytokine IL-6 | Before stimulation to Day 1 post stimulation
Cytokine IL-8 | Before stimulation to Day 1 post stimulation
Cytokine IL-10 | Before stimulation to Day 1 post stimulation
Cytokine TNF | Before stimulation to Day 1 post stimulation
C-Reactive Protein level | At days 2 and 3 post stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Ziekenhuis, Eindhoven, Netherlands